CLINICAL TRIAL: NCT04287452
Title: Canine-Assisted ANxiety Reduction IN Emergency Care IV (CANINE IV)
Brief Title: Canine-Assisted ANxiety Reduction IN Emergency Care IV
Acronym: CANINE IV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been withdrawn due to the pandemic and lack of funding.
Sponsor: Indiana University (Other)
Collaborators: Healthcare Initiatives, Inc. (Unknown)
Responsible Party: Principal Investigator, Nicholas Pettit, Assistant Professor of Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001968358
Record Dates: First submitted 2020-02-12; First posted 2020-02-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Anxiety Acute; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Emergency department patients enrolled in the control arm will receive usual care. Emergency department providers enrolled in the control arm will work their shift as usual.
  Interventions: Other: Control
- Intervention (Active Comparator): Emergency department patients and providers in the intervention arm will be exposed to and/or interact with a certified therapy dog and handler
  Interventions: Other: Dog Therapy

INTERVENTIONS:
Other: Control — Control
  Arms: Control
Other: Dog Therapy — Exposure to certified therapy dogs and their handler.
  Arms: Intervention

SUMMARY:
Prior literature demonstrates that human stress can be reduced with exposure to animals. This study challenges current dogma by introducing a widely available, low cost method of dog therapy to reduce patient and provider stress. The objectives of this study are to determine if interaction with a certified therapy dog and handler can;

* decrease reported anxiety levels in emergency department (ED) patients,
* decrease salivary cortisol in ED patients,
* decrease total morphine equivalent dosing in the emergency department or at discharge and/or,
* decrease reported stress levels in emergency department providers caring for participating patients

when compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Age 18-89 years
* Chronic pain, defined as pain on most days for >6 weeks
* Triage pain score >6 out of 10

OR

* Age 18-89 years
* Currently experience crisis, including suicidality, or
* Meet the standard of a provider assessment of "severe stress" defined by their identification that the patient meets a score of greater than six on the FACES stress scale

Providers

• Faculty, residents, advanced practitioners, and nurses who work in the ED and identify themselves as being the nurse or physician of record for the enrolled patients.

Therapy Dog Handlers

• Handler of a certified therapy dog and volunteer of Eskenazi's Therapy Dog Program

Exclusion Criteria:

Patients

* Violent behavior
* Overt intoxication
* Non-English speaking
* Any reported prior fear or adverse reaction to dogs

Providers

• Any reported prior fear or adverse reaction to dogs

Therapy Dog Handlers

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalent narcotic administration in emergency department patients with chronic pain | Date of enrollment until emergency department discharge, up to 72 hours
  Total morphine equivalent narcotic administration while in the emergency department or as a discharge prescription will be recorded for enrolled patients.
Change in reported stress levels in ED patients with chronic pain using Wong-Baker FACES Scale (10 = worst) | Baseline and T1 (~45 minutes after baseline)
  Change in self reported stress levels of emergency department patients using a Wong-Baker FACES Scale for anxiety between baseline and T1
Change in salivary cortisol in ED patients with chronic pain | Baseline and T1 (~45 minutes after baseline)
  Change in salivary cortisol levels in emergency department patients between baseline and T1
Number of narcotic, sedative and/or neuroleptic doses administered in ED patients with emotional crisis | Date of enrollment until emergency department discharge, up to 72 hours
  Number of narcotic, sedative and/or neuroleptic doses administered in ED patients with emotional crisis
Change in reported stress levels in ED patients with emotional crisis using Wong-Baker FACES Scale (10 = worst) | Baseline and T1 (~45 minutes after baseline)
  Change in self reported stress levels of emergency department patients using a Wong-Baker FACES Scale for anxiety between baseline and T1
Change in salivary cortisol in ED patients with emotional crisis | Baseline and T1 (~45 minutes after baseline)
  Change in salivary cortisol levels in emergency department patients between baseline and T1

SECONDARY OUTCOMES:
Change in salivary cortisol levels in emergency department patients | Baseline and T1 (~45 minutes after baseline)
  Change in salivary cortisol levels in emergency department patients between baseline and T1

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi Health System, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun C, Stangler T, Narveson J, Pettingell S. Animal-assisted therapy as a pain relief intervention for children. Complement Ther Clin Pract. 2009 May;15(2):105-9. doi: 10.1016/j.ctcp.2009.02.008. Epub 2009 Mar 3. PMID 19341990
- [Background] Marcus DA, Bernstein CD, Constantin JM, Kunkel FA, Breuer P, Hanlon RB. Impact of animal-assisted therapy for outpatients with fibromyalgia. Pain Med. 2013 Jan;14(1):43-51. doi: 10.1111/j.1526-4637.2012.01522.x. Epub 2012 Nov 21. PMID 23170993
- [Background] Barker SB, Dawson KS. The effects of animal-assisted therapy on anxiety ratings of hospitalized psychiatric patients. Psychiatr Serv. 1998 Jun;49(6):797-801. doi: 10.1176/ps.49.6.797. PMID 9634160
- [Background] Munoz Lasa S, Maximo Bocanegra N, Valero Alcaide R, Atin Arratibel MA, Varela Donoso E, Ferriero G. Animal assisted interventions in neurorehabilitation: a review of the most recent literature. Neurologia. 2015 Jan-Feb;30(1):1-7. doi: 10.1016/j.nrl.2013.01.012. Epub 2013 May 1. English, Spanish. PMID 23642347
- [Background] Havey J, Vlasses F, Vlasses P, Ludwig P, Hackbarth D. The Effect of Animal-Assisted Therapy on Pain Medication Use After Joint Replacement. Anthrozoos 2014; 27: 361-369.
- [Background] Smith DD, Kellar J, Walters EL, Reibling ET, Phan T, Green SM. Does emergency physician empathy reduce thoughts of litigation? A randomised trial. Emerg Med J. 2016 Aug;33(8):548-52. doi: 10.1136/emermed-2015-205312. Epub 2016 Mar 21. PMID 27002161
- [Background] Kelm Z, Womer J, Walter JK, Feudtner C. Interventions to cultivate physician empathy: a systematic review. BMC Med Educ. 2014 Oct 14;14:219. doi: 10.1186/1472-6920-14-219. PMID 25315848